CLINICAL TRIAL: NCT04800913
Title: The Role of Multimodality Imaging in Left Atrial Appendage Closure
Acronym: MILAAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hungarian Institute of Cardiology (Other Government)
Responsible Party: Principal Investigator, Anita Zadori MD, PhD, cardiologist, Hungarian Institute of Cardiology (Gottsegen National Cardiovascular Center), Hungarian Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MILAAC
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ischemic stroke; left atrial appendage closure; bleeding
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Hemorrhage | interventions — Multimodal Imaging

STUDY DESIGN:
Intervention Model Description: Prospective randomized one-centre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Multimodal imaging (Experimental): Preoperative 2D/3D TOE AND MDCT for appendage characterisation and sizing
  Operative 2D/3D TOE and fluoroscopy/angiography for guiding and checking the procedural events and success
  Postoperative 2D/3D TOE and MDCT to assess the complications (peri-device leak, thrombus)
  Interventions: Diagnostic Test: Multimodal imaging
- Standard imaging (Experimental): Preoperative MDCT for appendage characterisation and sizing
  Operative 2D/3D TOE and fluoroscopy/angiography for guiding and checking the procedural events and success
  Postoperative 2D/3D TOE and MDCT to assess the complications (peri-device leak, thrombus)
  Interventions: Diagnostic Test: Standard imaging

INTERVENTIONS:
Diagnostic Test: Multimodal imaging — Preoperative 2D/3D TOE and MDCT, operative 2D/3D TOE and fluoroscopy/angiography, postoperative 2D/3D TOE and MDCT
  Arms: Multimodal imaging
Diagnostic Test: Standard imaging — Preoperative MDCT, operative 2D/3D TOE and fluoroscopy/angiography, postoperative 2D/3D TOE and MDCT
  Arms: Standard imaging

SUMMARY:
The aim of the present prospective, randomized single-centre study is to examine the success rate, safety, overall preoperative and operative burden and long-time outcome of percutaneous left atrial appendage closure procedures after unimodal and multimodal preprocedural imaging.

According to the investigators' primary hypothesis, simple, unimodal preprocedural imaging does not increase procedural burden of LAAC (total radiation dose, procedure time, fluoroscopy time, contrast amount). The investigators assume, that the success rate and safety of LAAC procedures is not reduced using unimodal preoperative imaging.

Regarding to postoperative imaging, the investigators aim to compare the sensitivity of different imaging techniques in detecting postoperative complications. We assume, that multimodal imaging technique increases the accuracy and sensitivity of the detection of postoperative complications (PDL, device thrombi).

DETAILED DESCRIPTION:
Left atrial appendage closure (LAAC) is an increasingly used non-pharmacologic strategy to prevent stroke in patients with atrial fibrillation who have absolute or relative contraindications to long-term oral anticoagulant therapy, mainly due to previous major bleeding or high bleeding risk. As the majority of candidates are elderly patients with multiple morbidities, the reduction of procedural burden is of huge significance.

The aim of the present prospective, randomized, single-centre study is to examine the non-inferiority of unimodal (MDCT) vs. multimodal (MDCT+TOE) preprocedural imaging in percutaneous left atrial appendage closure. The investigators are going to assess the success rate, safety and complications of LAAC procedures, and determine the procedural burden (total radiation dose, procedure time, fluoroscopy time, contrast amount) of the interventions after preprocedural unimodal and multimodal appendage characterization and device sizing. Multimodal procedural guidance (2D/3D TOE, fluoroscopy-angiography) and multimodal postprocedural imaging (2D/3D TOE, MDCT) is going to be used to identify complications (peri-device leak, thrombus). The investigators are planning to compare the accuracy and additive value of different postoperative imaging techniques.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who have clinical indication to LAAC and are undergoing percutaneous LAAC procedure in Gottsegen National Cardiovascular Center from 10.03.2021 to 31.12.2025
* Age above 18 years
* Informed consent
* Legal capacity

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Incapacitation
* Absence of consent
* Esophageal stenosis or diverticulum
* Active esophageal bleeding
* CT-contrast agent allergy
* Severe chronic kidney disease (GFR<15 ml/min/1,73 m2)
* Appendage thrombus (mobile/with significant embolic risk)
* Life expectancy shorter than 12 months
* Active infection
* Significant mitral valve stenosis
* Mechanical heart valve
* Open heart surgery is indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Effective radiation dose | Periprocedural (1 month) interval
  Total radiation dose of the patient resorbed during LAAC imaging and intervention (mSv)

SECONDARY OUTCOMES:
Fluoroscopy time | during the procedure
  during LAAC procedure (min)
Procedure time | during the procedure
  of LAAC procedure (min)
Contrast media amount | during the procedure
  used during LAAC procedure (ml)
Rate of successful implantations | during the procedure
  left atrial appendage occluder successfully deployed and released
Rate of patients with adequate seal of closure device | 6 weeks post-procedure
  Adequate seal defined as no leak or residual leak< 5 mm established by postoperative TOE
Rate of procedural complications | within 30 days post-procedure
  Thromboembolic events, myocardial infarction, bleeding events, vascular complications, pericardial effusion, tamponade, infections, allergic reactions, renal insufficiency, device/air embolism, mortality
Rate of clinical events | 2 years post-procedure
  Composite endpoint of thromboembolic events (ischemic stroke, TIA, systemic embolism)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Zadori, MD, PhD, Principal Investigator — 0036303837011, anita.zadori@gokvi.hu
Locations (1):
- Hungarian Institute of Cardiology (Gottsegen National Cardiovascular Center), Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Reddy VY, Doshi SK, Kar S, Gibson DN, Price MJ, Huber K, Horton RP, Buchbinder M, Neuzil P, Gordon NT, Holmes DR Jr; PREVAIL and PROTECT AF Investigators. 5-Year Outcomes After Left Atrial Appendage Closure: From the PREVAIL and PROTECT AF Trials. J Am Coll Cardiol. 2017 Dec 19;70(24):2964-2975. doi: 10.1016/j.jacc.2017.10.021. Epub 2017 Nov 4. PMID 29103847
- [Background] Osmancik P, Tousek P, Herman D, Neuzil P, Hala P, Stasek J, Haman L, Kala P, Poloczek M, Branny M, Chovancik J, Cervinka P, Holy J, Vancura V, Rokyta R, Taborsky M, Kovarnik T, Zemanek D, Peichl P, Haskova S, Jarkovsky J, Widimsky P; PRAGUE-17 Investigators. Interventional left atrial appendage closure vs novel anticoagulation agents in patients with atrial fibrillation indicated for long-term anticoagulation (PRAGUE-17 study). Am Heart J. 2017 Jan;183:108-114. doi: 10.1016/j.ahj.2016.10.003. Epub 2016 Oct 11. PMID 27979034
- [Background] Nucifora G, Faletra FF, Regoli F, Pasotti E, Pedrazzini G, Moccetti T, Auricchio A. Evaluation of the left atrial appendage with real-time 3-dimensional transesophageal echocardiography: implications for catheter-based left atrial appendage closure. Circ Cardiovasc Imaging. 2011 Sep;4(5):514-23. doi: 10.1161/CIRCIMAGING.111.963892. Epub 2011 Jul 7. PMID 21737601
- [Background] Rajwani A, Nelson AJ, Shirazi MG, Disney PJS, Teo KSL, Wong DTL, Young GD, Worthley SG. CT sizing for left atrial appendage closure is associated with favourable outcomes for procedural safety. Eur Heart J Cardiovasc Imaging. 2017 Dec 1;18(12):1361-1368. doi: 10.1093/ehjci/jew212. PMID 28013284
- [Background] Sievert H, Lesh MD, Trepels T, Omran H, Bartorelli A, Della Bella P, Nakai T, Reisman M, DiMario C, Block P, Kramer P, Fleschenberg D, Krumsdorf U, Scherer D. Percutaneous left atrial appendage transcatheter occlusion to prevent stroke in high-risk patients with atrial fibrillation: early clinical experience. Circulation. 2002 Apr 23;105(16):1887-9. doi: 10.1161/01.cir.0000015698.54752.6d. PMID 11997272
- [Background] Qamar SR, Jalal S, Nicolaou S, Tsang M, Gilhofer T, Saw J. Comparison of cardiac computed tomography angiography and transoesophageal echocardiography for device surveillance after left atrial appendage closure. EuroIntervention. 2019 Oct 20;15(8):663-670. doi: 10.4244/EIJ-D-18-01107. PMID 31217149